CLINICAL TRIAL: NCT06503497
Title: A Single-center, Single-arm, Open-label, Dose-escalation Clinical Study to Evaluate the Safety and Anti-tumor Efficacy of Second-line Systemic Chemotherapy Sequential NKG2D CAR-NK Cell Therapy for Pancreatic Cancer
Brief Title: A Trail of Second-line Chemotherapy Sequential NKG2D CAR-NK Cell Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-C1/22A1-08-B
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-07

CONDITIONS: Pancreatic Cancer Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy Sequential NKG2D CAR-NK Cell (Experimental)
  Interventions: Biological: chemotherapy sequential CAR-NK cell infusion

INTERVENTIONS:
Biological: chemotherapy sequential CAR-NK cell infusion — In each chemotherapy cycle, patients received 2 intravenous infusions of CAR-NK on days 2 and 3 after each chemotherapy was discontinued.

SUMMARY:
This is a single-center, single-arm, open-label, dose-escalation clinical study to evaluate the safety and anti-tumor efficacy of second-line systemic chemotherapy sequential NKG2D CAR-NK cell therapy for pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18~75 years old (including boundary value), both male and female.
* 2. Histologically or cytologically confirmed pancreatic ductal adenocarcinoma or IPMN carcinosis with at least first-line systemic therapy failure.
* 3. Zubrod-ECOG-WHO score (see Annex 2) on a scale of 0-2.
* 4. Life expectancy of at least 3 months at screening, as judged by the investigator.
* 5. At least one stably evaluable target lesion according to RECIST1.1 criteria.
* 6. Subject has adequate organ and bone marrow function. Laboratory screening results should be within the stable range described below, with no ongoing supportive care ("yellowing" therapy such as PTCD, ENBD, or bile duct stenting is allowed when pancreatic cancer invades the common bile duct).
* 7. Remission of all toxicities due to prior antineoplastic therapy to Grade 0~1 (according to NCI CTCAE version 5.0) or to acceptable levels for inclusion/exclusion criteria.
* 8. Childbearing status: not pregnant, and if of childbearing potential, willing to use effective contraception from the time of signing the informed consent form to 6 months after the last cell infusion (females of childbearing potential include premenopausal females and females within 2 years of postmenopause).
* 9. Subjects must sign and date written informed consent.
* 10. Subjects must be voluntary and able to comply with predetermined treatment regimens, laboratory tests, follow-up, and other study requirements.

Exclusion Criteria:

* 1. Pregnant and lactating females.
* 2. Positive serology for HIV, Treponema pallidum or HCV (those who are HCV antibody positive but HCV-RNA negative, stable syphilis and inactive patients can be included).
* 3. Any active infection, including but not limited to active tuberculosis, HBV infection (including HBsAg positive, or HBcAb positive with HBV DNA above the lower limit of laboratory testing), Epstein-Barr virus (EBV) DNA positive, cytomegalovirus (CMV) DNA positive or novel coronavirus (new coronavirus) nucleic acid positive, and other bacterial, viral, or fungal infections requiring drug treatment;
* 4. History of malignancy within 5 years, with the exception of basal cell carcinoma of the skin and carcinoma in situ of the cervix.
* 5. Any other health condition that, in the judgment of the investigator, would preclude participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | within 28 days after NKG2D CAR-NK treatment
  Determine the optimal agent for NKG2D CAR-NK at maximum tolerated dose
Dose limiting toxicity | From enrollment of the first subject to completion of follow-up of the last subject up to 2 years
  Describe the adverse events of limiting further increases in the dose of NKG2D CAR-NK

SECONDARY OUTCOMES:
Effectiveness evaluation | At weeks 4、8 and months 3、6、9、12、16、20 and 24 after treatment
  Objective Response Rate (ORR) According to Response Evaluation Criteria In Solid Tumors Version 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- the first affiliated hospital of Zhejiang University，school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No